CLINICAL TRIAL: NCT01911988
Title: Study of Association Between Peripheral Immune Cells and Recurrence in Stage II/III Colorectal Cancer
Acronym: PICC-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Long Cui, Director, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHGC 001
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer
Keywords: Peripheral immune cells; Colorectal Cancers; Stage II/ Stage III; Recurrence; Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colon&Rectal Stage II /Stage III

SUMMARY:
The purpose of this study is to determine association between Peripheral Immune Cells(PIC) and recurrence in stage II/III colorectal cancer

DETAILED DESCRIPTION:
The investigators hypothesize differentiation of Peripheral Immune Cells(PIC) would result in resistance of chemotherapy and tumor local of metastatic recurrence.

The primary endpoint of this study is Disease Free Survival and the secondary endpoint is 5-year Overall Survival.

5ml peripheral blood will be sorted and counted through flow cytometry at the point of before primary treatment(surgery for colon cancers, neoadjuvant therapy for rectal cancers) , before the first chemotherapy postoperatively and 1 month after last chemotherapy.

Patients will be followed up with 3 monthly assessments in the first two years and 6 monthly assessments in the rest three years. Stratification factors include age , BMI , gender , tumor location , rectal or colon cancer stage,the chemotherapy (FOLFOX, XELOX, DeGramont or Capecitabine ),laparoscopic or laprotomy, anastomosis, concomitant medications and complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinically /Pahohistologically diagnosed as stageII/III CRC
* ECOG 0-2
* Age 18-90
* Gender both

Exclusion Criteria:

* Distant metastases noticed before or during surgery
* History of malignant tumor disease
* History of autoimmune diseases or immunodeficiencies
* History of hematological disease
* History of hepatic cirrhosis or Splenomegaly
* History of chronic kidney disease
* History of organ transplant
* History of chronic inflammatory disease
* Use of hematological drugs within 1 year prior to surgery
* Use of immunodulatory drugs within 1 year prior to surgery
* Use of chemotherapeutic drugs within 1 year prior to surgery
* Long term Use of non-steroid anti-inflammatory drugs(>6 months)
* Unable or Unwilling to undergo all the standard treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II /Stage III Colorectal Patients
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2013-06; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  The time from resection to the time of disease recurrence(local or metastatic) or death from any cause.

SECONDARY OUTCOMES:
5 years overall survival | 5 years or the time of death
  the time from resection to the time of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Long Cui, MD, PhD, Study Chair — Medical Center of Colon&Rectal Cancers, Shanghai Xinhua Hospital affiliated to Shanghai Jiaotong University
Locations (1):
- Medical Center of Colon&Rectal Cancers, Shanghai, China